CLINICAL TRIAL: NCT04947202
Title: Observational, Retrospective, Multi-center Clinical Study on the Safety of SAFIL® MESH in Patients Undergoing Reinforcement of Soft Tissues After Abdominal Wall Surgery or Other Fascial Defects
Brief Title: Clinical Study on the Safety of SAFIL® MESH
Acronym: SAFIL_MESH
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2040
Record Dates: First submitted 2021-06-16; First posted 2021-07-01 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Abdominal Wall Defect; Ventral Hernia; Abdominal Hernia; Fascial Hernia
Keywords: Reinforcement of Soft Tissues; Hernioplasty; mesh repair
MeSH Terms: conditions — Hernia, Ventral; Hernia, Abdominal | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Safil Mesh
  Interventions: Device: Hernioplasty

INTERVENTIONS:
Device: Hernioplasty — Hernioplasty is the repair of the defect using mesh patches.

SUMMARY:
Observational, Retrospective, Multi-center Clinical Study on the Safety of SAFIL® MESH in Patients Undergoing Reinforcement of Soft Tissues After Abdominal Wall Surgery or Other Fascial Defects

DETAILED DESCRIPTION:
The study design is a retrospective case-note series of patients that have undergone reinforcement of soft tissues with Safil® Mesh after abdominal wall surgery or other fascial defects between the period January 2019 - November 2020

ELIGIBILITY:
Inclusion Criteria:

* Patients operated between January 2019 - November 2020 for abdominal wall surgery or other fascial defects and received Safil® Mesh

Exclusion Criteria:

* No exclusion criteria have been set.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated between January 2019 - November 2020 for abdominal wall surgery or other fascial defects and received Safil® Mesh
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Hernia rate | at one follow-up 12-30 months after initial intervention
  Rate of hernias occuring during follow-up of retrospectively included patients

SECONDARY OUTCOMES:
Intra-operative complications | intraoperatively
  Retrospective documentation of Number of Participants with intraoperative Complications
Post-operative complications | at one follow-up 12-30 months after initial intervention
  Number of retrospectively included participants having complications during follow-up of
Reintervention rate | at one follow-up 12-30 months after initial intervention
  Complications leading to reintervention during follow-up of retrospectively included patients

OTHER OUTCOMES:
Demographic data of the patient: age | preoperatively
  Retrospective documentation of Demographic data of the patient for descriptive purposes: age of patients at time of surgery
Demographic data of the patient: sex | preoperatively
  Retrospective documentation of Demographic data of the patient for descriptive purposes: sex
Demographic data of the patient: weight | preoperatively
  Retrospective documentation of Demographic data of the patient for descriptive purposes: weight and height are documented to calculate body mass index
Demographic data of the patient: height | preoperatively
  Retrospective documentation of Demographic data of the patient for descriptive purposes: weight and height are documented to calculate body mass index
Demographic data of the patient: general health status | preoperatively
  Retrospective documentation of Demographic data of the patient for descriptive purposes: general health status according to ASA classification (ASA I: healthy patient; ASA II: A patient with mild systemic disease; ASA III: A patient with severe systemic disease; ASA IV: A patient with severe systemic disease that is a constant threat to life; ASA V: A moribund patient who is not expected to survive without the operation)
Demographic data of the patient: risk factors | preoperatively
  Retrospective documentation of Demographic data of the patient for descriptive purposes: risk factors (smoker, alcohol abuse, previous surgery of abdominal hernia, chronic immunosuppression, chronic cortison treatment, abdominal aortic aneurysm, anticoagulantic treatment)
Surgery details: Type of intervention | intraoperative
  Retrospective documentation of surgery details for descriptive purposes:
  Type of intervention (elective / emergency)
Surgery details: access | intraoperative
  Retrospective documentation of surgery details for descriptive purposes:
  access (open / laparoscopic / laparoscopic with conversion)
Surgery details: anesthetics | intraoperative
  Retrospective documentation of surgery details for descriptive purposes:
  anesthetics (general / regional / local)
Surgery details: duration of surgery | intraoperative
  Retrospective documentation of surgery details for descriptive purposes:
  duration of surgery
Surgery details: details on implanted mesh | intraoperative
  Retrospective documentation of surgery details for descriptive purposes:
  details on implanted mesh (number / sizes)
Surgery details: closure technology | intraoperative
  Retrospective documentation of surgery details for descriptive purposes:
  closure technology (absorbable suture, non absorbable suture, single-knot, continuous suture, adhesives)

CONTACTS AND LOCATIONS:
Overall Officials: Izaskun Badiola Bergara, Dr., Principal Investigator — Hospital Galdakao-Usansolo
Locations (2):
- Spain (2):
  - Hospital Galdakao-Usansolo, Galdakao, Bizkaia
  - Hospital Universitario de Salamanca, Salamanca